CLINICAL TRIAL: NCT02243774
Title: Mail Outreach To Increase Vaccination Acceptance Through Engagement
Acronym: MOTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Centers for Medicare and Medicaid Services (U.S. Federal Agency); United States Social and Behavioral Sciences Team (Unknown)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-P-001821
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Influenza, Human; Influenza; Human Flu
Keywords: Vaccination; Immunization; Randomized Controlled Trial; Prevention & Control; Preventive Measures; Health Promotion; Medicare; Intention Prompts; Letters
MeSH Terms: conditions — Influenza, Human

ARMS (5):
- No letter (No Intervention): Individuals randomized to the control group who will not receive any of the four letters
- Core letter signed by Surgeon General (Experimental): Individuals randomized to receive only a core letter signed by the Surgeon General
  Interventions: Behavioral: Core letter signed by Surgeon General
- Core letter signed by Director of the National Vaccine Program (Experimental): Individuals randomized to receive only a core letter signed by the Director of the National Vaccine Program
  Interventions: Behavioral: Core letter signed by the Director of the National Vaccine Program
- Core letter signed by Surgeon General + implementation prompt (Experimental): Individuals randomized to receive a core letter signed by the Surgeon General with an implementation intention prompt added in an appended P.S. tag region below the signature line
  Interventions: Behavioral: Core letter signed by Surgeon General + implementation prompt
- Core letter signed by SG + enhanced implementation prompt (Experimental): Individuals randomized to receive a core letter signed by the Surgeon General (SG) with an enhanced implementation intention prompt added in an appended P.S. tag region below the signature line
  Interventions: Behavioral: Core letter signed by SG + enhanced implementation prompt

INTERVENTIONS:
Behavioral: Core letter signed by Surgeon General — The core letter provides information about influenza and the risks associated with it, incorporating a number of behavioral insights. All four letters evaluated in this study will contain the same tops and bodies that are included in the core letter, but the signature and P.S. tag region will differ among the various intervention groups. In this intervention, the core letter is signed by and includes a picture of the Surgeon General. The letter ends after the signature line and the space beneath the signature line is left blank where a P.S. tag region could be appended.
  Arms: Core letter signed by Surgeon General
Behavioral: Core letter signed by the Director of the National Vaccine Program — The core letter is signed by and includes a picture of the Director of the National Vaccine Program. The letter ends after the signature line and the space beneath the signature line is left blank where a P.S. tag region could be appended.
  Arms: Core letter signed by Director of the National Vaccine Program
Behavioral: Core letter signed by Surgeon General + implementation prompt — The core letter is signed by and includes a picture of the Surgeon General. Below the signature line of the core letter, an implementation intention prompt is provided in the P.S. tag region that invites the recipient to write in the day of week, month, day, and time at which he or she plans to get vaccinated.
  Arms: Core letter signed by Surgeon General + implementation prompt
Behavioral: Core letter signed by SG + enhanced implementation prompt — The core letter is signed by and includes a picture of the Surgeon General (SG). Below the signature line of the core letter, an enhanced implementation intention prompt is provided in the P.S. tag region that prompts recipients to "decide now" - by checking one of two boxes - indicating they will or will not get vaccinated. The options use language that highlights the losses incumbent in refusing to vaccinate. In addition, an implementation intention prompt is embedded into the checkbox for indicating a choice to be vaccinated.
  Arms: Core letter signed by SG + enhanced implementation prompt

SUMMARY:
The aim of this study is to determine whether receiving a core letter signed by the Surgeon General or the Director of the National Vaccine Program that provides only information about influenza, or a core letter signed by the Surgeon General with an added basic or enhanced implementation prompt, will increase rates of influenza vaccination among Medicare beneficiaries when compared to a control group.

ELIGIBILITY:
Medicare fee-for-service beneficiaries aged 66 and older are eligible for study inclusion. There will be no additional exclusion criteria.

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 228000 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of study participants who receive influenza vaccination | 4 months
  Primary outcome of interest, determined from administrative claims data, will be the number of beneficiaries in each experimental group who receive an influenza vaccination between the date letter is mailed in September 2014 and January 31, 2015

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- Centers for Medicare & Medicaid Services, Baltimore, Maryland, United States